CLINICAL TRIAL: NCT04292327
Title: Clinical Progressive Characteristics and Treatment Effects of 2019-novel Coronavirus(2019-nCoV)
Brief Title: Clinical Progressive Characteristics and Treatment Effects of 2019-novel Coronavirus
Acronym: 2019-nCoV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, associate chief physician, Fujian Provincial Hospital
Other Study IDs: KY-2020-24.01
Record Dates: First submitted 2020-02-23; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Pneumonia Caused by Human Coronavirus
Keywords: 2019-novel coronavirus; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The ordinary COVID-19: Consistent with the diagnosis of ordinary COVID-19.
- The heavy COVID-19.: Consistent with the diagnosis of heavy COVID-19.
- The critical COVID-19: Consistent with the diagnosis of critical COVID-19

SUMMARY:
Objects: The purpose of this study was to observe the characteristics of morbidity, disease progression and therapeutic effects of 2019-novel coronavirus pneumonia patients with different clinical types.

Method: A single center, retrospective and observational study was used to collect COVID-19 patients admitted to Wuhan Infectious Diseases Hospital (Wuhan JinYinTan Hospital) from January 2020 to March 2020. The general information, first clinical symptoms, hospitalization days, laboratory examination, CT examination, antiviral drugs, immune enhancers, traditional Chinese medicine treatment and other clinical intervention measures were recorded, and the nutritional status and prognosis of the patients were recorded. confirm COVID-19 's disease progression, clinical characteristics, disease severity and treatment effects. To compare the characteristics of disease progression, clinical features, disease severity and therapeutic effect of different types of COVID-19.

Outcomes: The characteristics of disease progression, clinical features, disease severity and therapeutic effect of different types of COVID-19.

Conclusion: The characteristics of disease progression, clinical features and therapeutic effect of different types of COVID-19.

DETAILED DESCRIPTION:
Since December 2019, patients with unexplained pneumonia have appeared in some medical institutions in Wuhan, China. Nucleic acid testing was completed on January 10, 2020, which was confirmed to be caused by 2019-novel coronavirus. In 2020, the World Health Organization(WHO) named the virus 2019-novel coronavirus(2019-nCoV). The WHO announced that the pneumonia caused by 2019-nCoV is officially called COVID-19. Today, more than 70,000 cases have been confirmed and more than 2,000 patients have died.

At present, the epidemiological characteristics, laboratory indicators, imaging features and clinical treatment effects of COVID-19 should be reported, but the sample size is small. Large sample studies are still needed to further confirm COVID-19 's disease progression, clinical characteristics, disease severity and treatment effects, so as to provide a scientific basis for future clinical treatment. Therefore, it is particularly important to further review the relationship between the characteristics and prognosis of such patients.

ELIGIBILITY:
Inclusion criteria.

1. 2019-nCov (SARA-Cov-2) nucleic acid positive detected by PCR.
2. Older than 18 years old and younger than 75 years old.
3. Meet the diagnostic criteria of COVID-19 for different types (including ordinary type, heavy type and critical type)

Exclusion criteria.

1. the age is less than 18 years old;
2. pregnant or lactating women;
3. severe underlying diseases, such as advanced malignant tumor, end-stage lung disease, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collect COVID-19 patients admitted to Wuhan Infectious Diseases Hospital (Wuhan JinYinTan Hospital) from January 2020 to March 2020
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 day
  The mortality of COVID-19 in 28 days
The time interval of Nucleic acid detection become negative | 28 day
  The time interval of COVID-19 form nucleic acid confirmed to the nucleic acid detection turn into negative.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuling Shang, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided